CLINICAL TRIAL: NCT05855642
Title: The Accuracy And Safety of Trans Pedicular Screw Fixation of The Sub-axial Cervical Spine Using A Triad- Dependent Technique (TDT)
Brief Title: Accuracy And Safety of Trans Pedicular Screw Fixation of The Sub-axial Cervical Spine Using A Triad- Dependent Technique
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdelrahman Saleh El Attar, principal investigator, Assiut University
Other Study IDs: ASTPSF
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Pedicle Screw; CPS

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: All patients presented with degenerative or traumatic cervical spine matched the inclusion criteria will enrolled in our study from April 2023 to April 2024.

SUMMARY:
The use of the pedicle screw system has become increasingly popular for treating an unstable cervical spine resulting from traumatic, degenerative, inflammatory, and neoplastic conditions. Because the cervical pedicle screw (CPS) has superior bio mechanical stability as the lateral mass screw or trans articular screw , pedicle screws allow for shorter instrumentation with improved spinal alignment. However, CPS insertion is technically demanding because of the anatomical variations in cervical pedicle size, lack of anatomical landmarks, small pedicle diameter, and the large transverse angle of cervical pedicles . The potential risk of injury to neurovascular structures, such as the vertebral artery, spinal cord, or nerve roots, caused by CPS remains a great concern. Therefore, accurate and safe CPS insertion techniques are necessary.

DETAILED DESCRIPTION:
The use of the pedicle screw system has become increasingly popular for treating an unstable cervical spine resulting from traumatic, degenerative, inflammatory, and neoplastic conditions. Because the cervical pedicle screw (CPS) has superior bio mechanical stability as the lateral mass screw or trans articular screw , pedicle screws allow for shorter instrumentation with improved spinal alignment. However, CPS insertion is technically demanding because of the anatomical variations in cervical pedicle size, lack of anatomical landmarks, small pedicle diameter, and the large transverse angle of cervical pedicles . The potential risk of injury to neurovascular structures, such as the vertebral artery, spinal cord, or nerve roots, caused by CPS remains a great concern. Therefore, accurate and safe CPS insertion techniques are necessary.

Although a number of studies have evaluated the morphometric of cervical pedicles to support accurate placement of pedicle screws , the results are inconclusive. Therefore, several techniques using lateral fluoroscopy , pedicle axis view by oblique fluoroscopy , laminoframinotomy and computer-assisted navigation systems for CPS insertion have been advocated. Determining an appropriate entry point for screw insertion as well as a proper trajectory angle of the screw on the axial plane is important for successful pedicle screw placement. Here, we present our method using a fashioned triad- dependent technique (TDT) which is a combination of three methods 1-preoperative planning of the selected pedicle using 3-diamentional multi-slice CT to measure pedicle transverse angle (PTA) , pedicle outer diameter(POD)and pedicle trajectory -contralateral lamina angle 2-AP and oblique fluoroscopy to determine pedicle entry point (PEP), parallelism to vertebral end plate and 4 direction cortical violation (medial, lateral, superior, inferior) 3-interlaminar confirmatory key hole for tactile cue of medial ,superior, and inferior borders of the pedicle and related nerve root to evaluate the accuracy and safety of pedicle screw placement in patients with sub axial cervical spine disorders treated using our method.

ELIGIBILITY:
Inclusion Criteria:

1. traumatic sub axial cervical spine injuries.
2. degenerative cervical spine disorders necessitating cervical fusion

Exclusion Criteria:

1. congenital anomaly of the cervical spine
2. scoliotic deformity of the cervical spine
3. sever osteoporosis
4. congenital malformation of the pedicle.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All patients presented with degenerative or traumatic cervical spine matched the inclusion criteria will enrolled in our study from April 2023 to April 2024
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Radiological accuracy | Immediately post Operative
  A. X-ray AP and lateral
  B. MSCT: Placements of pedicle screws will be assessed using CT data and outcome-based classifications:
  2 mm increment classification:
  * Type 0 (good): Screw within the pedicle medullary canal.
  * Type 1 (acceptable): Minimal penetration of the pedicle wall by the screw (<2 mm of medial or lateral cortical perforation or anterior cortex perforation).
  * Type 2 (unacceptable): Less than half of the diameter of the screw was outside the pedicle wall (2-4 mm of perforation).
  * Type 3 (grievous): More than half of the diameter of the screw was outside the pedicle wall (>4 mm of perforation) (spinal cord injury or screw abutting vertebral artery).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotani Y, Cunningham BW, Abumi K, McAfee PC. Biomechanical analysis of cervical stabilization systems. An assessment of transpedicular screw fixation in the cervical spine. Spine (Phila Pa 1976). 1994 Nov 15;19(22):2529-39. doi: 10.1097/00007632-199411001-00007. PMID 7855677
- [Background] Jones EL, Heller JG, Silcox DH, Hutton WC. Cervical pedicle screws versus lateral mass screws. Anatomic feasibility and biomechanical comparison. Spine (Phila Pa 1976). 1997 May 1;22(9):977-82. doi: 10.1097/00007632-199705010-00009. PMID 9152447
- [Background] Karaikovic EE, Daubs MD, Madsen RW, Gaines RW Jr. Morphologic characteristics of human cervical pedicles. Spine (Phila Pa 1976). 1997 Mar 1;22(5):493-500. doi: 10.1097/00007632-199703010-00005. PMID 9076880
- [Background] Ludwig SC, Kramer DL, Vaccaro AR, Albert TJ. Transpedicle screw fixation of the cervical spine. Clin Orthop Relat Res. 1999 Feb;(359):77-88. doi: 10.1097/00003086-199902000-00009. PMID 10078131
- [Background] Bredow J, Beyer F, Oppermann J, Kraus B, Meyer C, Stein G, Eysel P, Koy T. A novel classification of screw placement accuracy in the cervical spine. Technol Health Care. 2016 Nov 14;24(6):919-925. doi: 10.3233/THC-161246. PMID 27497461
- [Background] Aoude AA, Fortin M, Figueiredo R, Jarzem P, Ouellet J, Weber MH. Methods to determine pedicle screw placement accuracy in spine surgery: a systematic review. Eur Spine J. 2015 May;24(5):990-1004. doi: 10.1007/s00586-015-3853-x. Epub 2015 Mar 7. PMID 25749690
- [Background] Jo DJ, Seo EM, Kim KT, Kim SM, Lee SH. Cervical pedicle screw insertion using the technique with direct exposure of the pedicle by laminoforaminotomy. J Korean Neurosurg Soc. 2012 Nov;52(5):459-65. doi: 10.3340/jkns.2012.52.5.459. Epub 2012 Nov 30. PMID 23323166
- [Background] Yukawa Y, Kato F, Ito K, Horie Y, Hida T, Nakashima H, Machino M. Placement and complications of cervical pedicle screws in 144 cervical trauma patients using pedicle axis view techniques by fluoroscope. Eur Spine J. 2009 Sep;18(9):1293-9. doi: 10.1007/s00586-009-1032-7. Epub 2009 Jun 2. PMID 19488794